CLINICAL TRIAL: NCT01825057
Title: Three Strategies for Implementing Motivational Interviewing on Medical Inpatient Units: See One, Do One, Order One
Brief Title: Three Strategies for Implementing Motivational Interviewing on Medical Inpatient Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Martino, Professor of Psychiatry, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01DA034243 (NIH)
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: See One; Do One; Order One
Keywords: implementation study; motivational interviewing; substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: In this three-arm parallel assignment, study-eligible and consented provider participants are randomized to one of three conditions (See One, Do One, or Order One) in which they receive their respective motivational interviewing training in parallel with provider participants assigned to the other conditions.
Who Masked: Participant
Masking Description: Research staff independently screen, assess and obtain consent from eligible substance using patients admitted to the general medical hospitalist service. Patients are included if they are assigned to a participating provider according to the hospital's usual clinical administrative procedures. Thus, patients followed the randomization condition of their assigned provider, but they do not know how their providers have been trained to deliver MI and the providers do not know which patients assigned to them have been enrolled in the study. This approach permits a naturalistic test of the providers' ability to identify and intervene using MI with patients who misuse substances without patients or research staff prompting providers to do so.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- See One (Active Comparator): Providers in See One only receive MI workshop training, giving them an opportunity to "see" the MI intervention and learn how to conduct it. The trainer encourages them to screen their patients for substance misuse and apply MI as indicated.
  Interventions: Behavioral: See One
- Do One (Experimental): Following workshop training, MI-trained CL clinicians directly supervise providers' live bedside provision of MI to patients twice before beginning the trial and once midstream. In addition, providers have the option to request additional live supervision from CL clinicians during the trial, consistent with the apprenticeship model.
  Interventions: Behavioral: Do One
- Order One (Experimental): Following the workshop, providers either administer MI themselves or "order" a MI for delivery by one of the MI-trained CL clinicians. Only providers in Order One can specifically request MI through a separate CL order in the electronic health record. The physicians or PAs directly place MI orders. Nurses contact physicians or PAs to place the MI order. The CL clinicians are trained in MI via a clinical trials training approach: 1) a 2-day skill-building workshop; 2) three post-workshop supervised practice cases based on review of audio recorded sessions; and 3) follow-up monthly group supervision to maintain and monitor the CL clinicians' MI practice. CL clinicians also learned supervisory practices to provide live supervision to providers in Do One.
  Interventions: Behavioral: Order One

INTERVENTIONS:
Behavioral: See One — A 1-day workshop conducted by a member of the Motivational Interviewing Network of Trainers (MINT), according to MINT recommendations, to build providers' skills needed to use MI with patients who misuse substances.
  Other Names: Workshop
  Arms: See One
Behavioral: Do One — A 1-day workshop conducted by a member of the Motivational Interviewing Network of Trainers (MINT), according to MINT recommendations, to build providers' skills needed to use MI with patients who misuse substances. Following the workshop training, providers conduct two motivational interviews bedside with patients under the supervision of one of the MI-trained CL clinicians, who subsequently give them performance feedback and coaching. Providers receive one more supervised practice case mid-trial. In addition, they can request additional supervision at any point during the trial.
  Other Names: Workshop plus live supervision
  Arms: Do One
Behavioral: Order One — A 1-day workshop conducted by a member of the Motivational Interviewing Network of Trainers (MINT), according to MINT recommendations, to build providers' skills needed to use MI with patients who misuse substances. Following the workshop, providers have the option to conduct MI with patients themselves or to "order" a MI for delivery by one of the MI-trained CL clinicians.
  Other Names: Workshop plus consultation-liaison service
  Arms: Order One

SUMMARY:
General medical hospitals provide care for a disproportionate share of patients who misuse substances. Motivational interviewing (MI) is a well-recognized, evidenced-based substance use treatment. However, it is unclear which implementation strategies lead to the efficient and proficient uptake of MI in general medical settings, such as medical inpatient units. Because medical providers have multiple practice demands and time constraints, new practices have the greatest chance of being implemented if they are simple and compatible with existing workflows and systems. Two widely used strategies to bring specialized practices into use within general hospital settings are the apprenticeship model of training and use of consultation-liaison (CL) services. The apprenticeship model requires that appropriate patients and trainers are available with high flexibility for teaching and supervision; when applied to behavioral counseling approaches, this model may be incompatible with the providers' medical role and time constraints. In contrast, ordering MI through CL is relatively simple, minimally burdensome, and highly compatible with the way clinicians secure other specialist services for their patients in the hospital. This cluster randomized controlled trial examines the effectiveness of three different strategies for integrating MI into the practice of medical providers working within an academically affiliated internal medicine hospitalist service. Specifically, the trial randomizes 38 healthcare providers to one of three conditions: (1) a continuing medical education workshop that provides background and "shows" healthcare providers how to conduct MI (the control condition, called SEE ONE); (2) a "see one, do one" apprenticeship model involving workshop training plus live supervision of bedside practice (DO ONE); and (3) ordering MI from CL after learning about it in a workshop (ORDER ONE). Following the respective MI trainings, each healthcare provider will be assessed for the provision of MI to 40 study-eligible inpatients, recruited by the research team after admission to our general medical units. Trial hypotheses are 1) the percentage of MI sessions delivered by providers to study-eligible inpatients will be higher in both Do One and Order One than See One, and 2) providers in both Do One and Order One will conduct MI sessions with greater integrity than those in See One. This study is an implementation trial examining provider, not patient, outcomes.

DETAILED DESCRIPTION:
General medical hospitals provide care for a disproportionate share of patients who abuse or are dependent upon substances. This group is among the most costly to treat and has the poorest medical and substance use outcomes. Motivational interviewing(MI) is a well-recognized, evidenced-based substance use treatment that has been adapted for use as a brief intervention in health care settings. MI is applicable to many health-related behavioral problems, and can be taught to a broad range of health care clinicians. However, it is unclear which implementation strategies will lead to the efficient and proficient uptake of MI in general medical settings, such as medical inpatient units.

Primary care clinicians have multiple practice demands and time constraints. New practices have the greatest chance of being implemented if they are simple and compatible with existing workflows and systems. Two widely used strategies to bring specialized practices into use within general hospital settings are the "see one, do one" apprenticeship model of training and use of consultation-liaison (CL) services. "See one, do one" has been a modus operandi in medical education for centuries and relies upon a competency-based supervision training approach. While it has been empirically validated in the specialty addiction field, less controlled testing of this implementation strategy is available in general medical settings. The apprenticeship approach requires that appropriate patients and trainers are available with high flexibility for teaching and supervision; when applied to behavioral counseling approaches, this may be seen as incompatible with the medical role and time constraints of clinicians. In contrast, ordering MI through CL is a relatively simple, minimally burdensome process and highly compatible with the way clinicians secure other specialist services for their patients in the hospital.

We propose to conduct a randomized controlled implementation trial using mixed quantitative and qualitative methods to examine the effectiveness of three different strategies for integrating MI into the practice of healthcare providers working within Yale New Haven Hospital's internal medicine hospitalist service and other general medical inpatient units. Specifically, we will randomize 40 healthcare providers to one of three conditions: (1) a continuing medical education workshop that provides background and "shows" healthcare providers how to conduct MI (the control condition, called SEE ONE); (2) a "see one, do one" apprenticeship model involving workshop training plus live supervision of bedside practice (DO ONE); and (3) ordering MI from CL after learning about it in a workshop (ORDER ONE). Following the respective MI trainings, each healthcare provider will be assessed for the provision of MI to 40 study-eligible inpatients, recruited by the research team after admission to our general medical units.We hypothesize that the percentage of MI sessions delivered by providers to study-eligible inpatients would be higher in both Do One and Order One than See One. We also hypothesize that providers in both Do One and Order One would conduct MI sessions with greater integrity (i.e., adherence to core components of MI and delivery of them with competence) than those in See One.

Please note, as an implementation trial, the primary outcomes for this study focus on provider behaviors, namely, uptake of MI sessions with patients and the adherence and competence in which they conduct MI sessions. No outcome data will be collected and reported at the patient level.

ELIGIBILITY:
For Healthcare provider participants:

Inclusion criteria :

* Assignment to one of the general medical inpatient units during day-time shifts; intensive care units will be excluded given the morbidity of patients in this setting.
* Volunteer to serve as study clinicians, attend a workshop about MI, and possibly receive live supervision.
* Agree to all procedures of this trial (randomization to training condition and of assigned patients, audio recording MI sessions, and completing assessments).

Exclusion criteria:

* Have been formally supervised to use MI with patients on the units.
* Intend to give notice that they plan to leave the hospital or are scheduled for medical or family leave such that they will not be able to interview 40 patients during the study period.

For patient participants:

Inclusion criteria:

* Are 18 years of age or older.
* Acknowledge use of a substance within past 28 days and meets screening criteria consistent with substance (illicit drugs, licit drugs that are used in a non-medically indicated fashion, alcohol, or nicotine) use disorder.
* Are willing to consent to audio recording of interview with the provider or CL clinician.

Exclusion criteria:

* Have an altered mental status such as delirium, encephalopathy, dementia or mental retardation or a score on the Confusion Assessment Method > 0 since this would impair provision of consent and ability to participate
* Inability to speak English. Most of providers are mono-lingual English speakers, and all MI integrity raters only speak English. We therefore do not have the capacity to include Spanish-only speaking patients in the study.
* Stroke (that precludes participation)
* Resides in a nursing home, skilled nursing facility or Hospice Care
* Receiving palliative care
* Deaf
* Unable to speak lucidly
* Previous participation in the protocol

An information sheet was requested and approved for a subset of patient subjects. This is due to the study being conducted within an acute medical inpatient unit, where conditions that might limit a person's ability to sign the consent form may occasionally occur. This subset of patients includes: patients that are physically unable to write (i.e. hand tremors, spinal cord injury, stroke that precludes signing, broken hand, broken shoulder, muscular dystrophy and other physical ailments preventing a patient from physically signing), unable to see (i.e. legally blind, uncontrolled type 2 diabetes mellitus which led to blurred vision), unable to read (i.e. patient does not have their glasses on them).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1211 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Martino, Ph.D., Principal Investigator — Yale University; Kimberly A Yonkers, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers upon request. PIs will screen requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon request, with review of request by Drs. Martino or Yonkers, beginning 10/24/19. Data requests will remain available for the subsequent 4 years.
Access Criteria: simply use the following emails for all data requests: steve.martino@yale.edu and kimberly.yonkers@yale.edu.

REFERENCES:
- [Background] Martino S, Zimbrean P, Forray A, Kaufman J, Desan P, Olmstead TA, Gueorguieva R, Howell H, McCaherty A, Yonkers KA. See One, Do One, Order One: a study protocol for cluster randomized controlled trial testing three strategies for implementing motivational interviewing on medical inpatient units. Implement Sci. 2015 Sep 29;10:138. doi: 10.1186/s13012-015-0327-9. PMID 26420671
- [Result] Martino S, Zimbrean P, Forray A, Kaufman JS, Desan PH, Olmstead TA, Gilstad-Hayden K, Gueorguieva R, Yonkers KA. Implementing Motivational Interviewing for Substance Misuse on Medical Inpatient Units: a Randomized Controlled Trial. J Gen Intern Med. 2019 Nov;34(11):2520-2529. doi: 10.1007/s11606-019-05257-3. Epub 2019 Aug 29. PMID 31468342
- [Derived] Serowik KL, Yonkers KA, Gilstad-Hayden K, Forray A, Zimbrean P, Martino S. Substance Use Disorder Detection Rates Among Providers of General Medical Inpatients. J Gen Intern Med. 2021 Mar;36(3):668-675. doi: 10.1007/s11606-020-06319-7. Epub 2020 Oct 27. PMID 33111239

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study's primary outcome and secondary outcomes are only collected and reported at the provider level - not at the patient level.
Period: Patient Study Flow
Arm/Group | See One | Do One | Order One
Started | 336 | 379 | 458
Completed | 336 | 379 | 458
Not Completed | 0 | 0 | 0
Period: Provider Study Flow
Arm/Group | See One | Do One | Order One
Started | 13 | 12 | 13
Completed | 13 | 12 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total provider and patient participant characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | See One | Do One | Order One | Total
Number analyzed (Participants) | 349 | 391 | 471 | 1211
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed in the rows represented are for two distinct participant groups in this study crossing the three conditions (See One, Do One, Order One), namely 38 providers and 1173 patients, which equals an overall number equal to 1211 participants.
  years
    Providers: number analyzed (Participants) | 13 | 12 | 13 | 38
    Providers | 39.2 (13.2) | 34.4 (8.9) | 32.2 (10.1) | 35.3 (11.0)
    Patients: number analyzed (Participants) | 336 | 379 | 458 | 1173
    Patients | 46.8 (14.0) | 46.3 (14.5) | 46.9 (14.5) | 46.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in the rows represented are for two distinct participant groups in this study crossing the three conditions (See One, Do One, Order One), namely 38 providers and 1173 patients, which equals an overall number equal to 1211 participants.
  Participants
    Providers: number analyzed (Participants) | 13 | 12 | 13 | 38
    Providers: Female | 11 | 10 | 12 | 33
    Providers: Male | 2 | 2 | 1 | 5
    Patients: number analyzed (Participants) | 336 | 379 | 458 | 1173
    Patients: Female | 152 | 182 | 200 | 534
    Patients: Male | 184 | 197 | 258 | 639
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number analyzed in the rows represented are for two distinct participant groups in this study crossing the three conditions (See One, Do One, Order One), namely 38 providers and 1173 patients, which equals an overall number equal to 1211 participants.
  Participants
    Providers: number analyzed (Participants) | 13 | 12 | 13 | 38
    Providers: non-Hispanic White | 10 | 11 | 8 | 29
    Providers: non-Hispanic African American | 1 | 1 | 1 | 3
    Providers: non-Hispanic Asian | 2 | 0 | 1 | 3
    Providers: Hispanic White | 0 | 0 | 2 | 2
    Providers: non-Hispanic Other Race | 0 | 0 | 1 | 1
    Patients: number analyzed (Participants) | 336 | 379 | 458 | 1173
    Patients: non-Hispanic White | 193 | 224 | 249 | 666
    Patients: non-Hispanic African American | 98 | 105 | 149 | 352
    Patients: non-Hispanic Asian | 0 | 0 | 0 | 0
    Patients: Hispanic White | 44 | 47 | 53 | 144
    Patients: non-Hispanic Other Race | 1 | 3 | 7 | 11
Type of provider [Count of Participants; unit: Participants] — Population: This baseline data was only collected for provider participants. Patient participants are not included.
  Participants
    number analyzed (Participants) | 13 | 12 | 13 | 38
    Registered Nurse | 6 | 6 | 7 | 19
    Physician's Assistant | 5 | 4 | 5 | 14
    Medical Doctor | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Motivation Interviewing Sessions Audio Recorded
Description: The percentage of audio recorded Motivational Interviewing sessions conducted by providers for their 40 consecutively enrolled study-eligible patients
Time Frame: Provider participants will be followed for the duration of the trial period, an expected average of 24 weeks to see 40 study-enrolled patients per provider.
Population: A percentage of MI sessions audio recorded was calculated for each provider, and a mean percentage was calculated by group.
Measure: Mean (Standard Deviation); unit: percentage of MI sessions audio recorded
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
percentage of MI sessions audio recorded | 0.8 (2.3) | 3.0 (5.4) | 20.5 (17.9)
Statistical Analysis 1: Comparison: Do One vs Order One; Test type: Superiority; p = 0.0009, Kruskal-Wallis — adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner Method; degrees of freedom = 2; Mean Difference (Final Values) = 17.5 — mean difference = Order One - Do One
Statistical Analysis 2: Comparison: See One vs Order One; Test type: Superiority; p < 0.0001, Kruskal-Wallis — Adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner Method; degrees of freedom = 2; Median Difference (Final Values) = 19.7 — mean difference = Order One - See One
Statistical Analysis 3: Comparison: See One vs Do One; Test type: Superiority; p = 0.4983, Kruskal-Wallis; degrees of freedom = 2; Mean Difference (Final Values) = 2.178 — mean difference = Do One - See One

2. Secondary Outcome: The Independent Tape Rater Scale - Fundamental Adherence Score
Description: The Independent Tape Rater Scale assessed the integrity of MI interviews. The Independent Tape Rater Scale includes 5 fundamental MI items important for building rapport and understanding patients' experiences (e.g. reflections), rated for adherence (i.e. the extent/frequency of intervention delivery) on a scale from 1 (not at all) to 7 (extensively). The fundamental adherence score is the average of these 5 items, with scores ranging from 1-7 and higher scores indicating greater adherence. Only MI sessions conducted within each study arm by the providers with patient participants were included in this analysis. Since 3 MI sessions were conducted by providers in See One, 11 sessions were conducted by providers in Do One, and 100 sessions were conducted by providers in Order One, this analysis includes 114 MI sessions as the unit of analysis.
Time Frame: All sessions conducted and recorded by providers with study-enrolled patients during the trial period, an expected 24 weeks per provider.
Population: Analysis sample includes the N=114 MI sessions completed by providers with study-enrolled patients across all training groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: MI Sessions completed by providers
Groups:
- See One: Providers in See One only received the workshop training, giving them an opportunity to "see" the MI intervention and learn how to conduct it. The trainer encouraged them to screen their patients for substance misuse and apply MI as indicated.
- Do One: Following workshop training, the MI-trained consultation-liaison clinicians directly supervised providers' live bedside provision of MI to patients twice before beginning the trial and once mid-trial. In addition, providers had the option to request additional live supervision from consultation-liaison clinicians during the trial, consistent with the apprenticeship model.
- Order One: Following the workshop training, providers had the option to either administer MI themselves or "order" a MI for delivery by one of the four MI-trained consultation-liaison clinicians.
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
Number analyzed (MI Sessions completed by providers) | 3 | 11 | 100
score on a scale | 4.00 (0.35) | 4.60 (0.80) | 5.22 (0.58)
Statistical Analysis 1: Comparison: Do One vs Order One; Test type: Superiority; p = 0.0217, Kruskal-Wallis — Adjusted for multiple comparisons using the Dwass, Steel, Critchlow-Fligner Method; Mean Difference (Final Values) = 0.62 — Mean difference = Order One - Do One
Statistical Analysis 2: Comparison: See One vs Order One; Test type: Superiority — mean difference is Order One - See One; p = 0.0126, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 1.22
Statistical Analysis 3: Comparison: See One vs Do One; Test type: Superiority; p = 0.4231, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.6 — mean difference is Do One - See One

3. Secondary Outcome: The Independent Tape Rater Scale- Fundamental Competence Score
Description: The Independent Tape Rater Scale assessed the integrity of MI interviews. The Independent Tape Rater Scale includes 5 fundamental MI items important for building rapport and understanding patients' experiences (e.g. reflections), rated for competency (i.e., the skill/quality of intervention delivery) on a scale of 1 (not at all) to 7 (excellent). The fundamental competence score is the average of these 5 items, for which there was adherence, with higher scores indicating greater competence. Only MI sessions conducted within each study arm by the providers with patient participants were included in this analysis. Since 3 MI sessions were conducted by providers in See One, 11 sessions were conducted by providers in Do One, and 100 sessions were conducted by providers in Order One, this analysis includes 114 MI sessions as the unit of analysis.
Time Frame: as for outcome 2
Population: Analysis population includes the N=114 MI sessions that were completed by providers across all training groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: MI Sessions completed by providers
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
Number analyzed (MI Sessions completed by providers) | 3 | 11 | 100
score on a scale | 3.67 (0.61) | 4.27 (0.43) | 4.71 (0.45)
Statistical Analysis 1: Comparison: Do One vs Order One; Test type: Superiority; p = 0.0091, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.44 — Mean difference = Order One - Do One
Statistical Analysis 2: Comparison: See One vs Order One; Test type: Superiority; p = 0.0196, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 1.04 — mean difference = Order One - See One
Statistical Analysis 3: Comparison: See One vs Do One; Test type: Superiority; p = 0.2832, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.60 — mean difference = Do One - See One

4. Secondary Outcome: The Independent Tape Rater Scale- Advanced Adherence Score
Description: The advanced adherence score is the average of these 5 items. The Independent Tape Rater Scale assessed the integrity of MI interviews. The Independent Tape Rater Scale includes 5 advanced MI items critical for eliciting patients' motivations for change (e.g., asking for reasons for change), rated for adherence (i.e., the extent/frequency of intervention delivery) on a scale of 1 (not at all) to 7 (extensively). The advanced adherence score is the average of these 5 items, with scores ranging from 1-7 and higher scores indicating greater adherence. Only MI sessions conducted within each study arm by the providers with patient participants were included in this analysis. Since 3 MI sessions were conducted by providers in See One, 11 sessions were conducted by providers in Do One, and 100 sessions were conducted by providers in Order One, this analysis includes 114 MI sessions as the unit of analysis.
Time Frame: as for outcome 2
Population: Analysis population includes the N=114 MI sessions that were completed by providers across all training groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: MI Sessions completed by providers
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
Number analyzed (MI Sessions completed by providers) | 3 | 11 | 100
score on a scale | 3.93 (0.58) | 4.38 (0.95) | 4.81 (0.65)
Statistical Analysis 1: Comparison: Do One vs Order One; Test type: Superiority; p = 0.1566, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.43 — Mean difference = Order One - Do One
Statistical Analysis 2: Comparison: See One vs Order One; Test type: Superiority; p = 0.0982, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.88 — mean difference = Order One - See One
Statistical Analysis 3: Comparison: See One vs Do One; Test type: Superiority; p = 0.6631, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.45 — mean difference = Do One - See One

5. Secondary Outcome: The Independent Tape Rater Scale- Advanced Competence Score
Description: The Independent Tape Rater Scale assessed the integrity of MI interviews. The Independent Tape Rater Scale includes 5 advanced MI items critical for eliciting patients' motivations for change (e.g., asking for reasons for change), rated for competency (i.e., the skill/quality of intervention delivery) on a scale of 1 (not at all) to 7 (excellent). The advanced competence score is the average of these 5 items, for which there was adherence, with higher scores indicating greater competence. Only MI sessions conducted within each study arm by the providers with patient participants were included in this analysis. Since 3 MI sessions were conducted by providers in See One, 11 sessions were conducted by providers in Do One, and 100 sessions were conducted by providers in Order One, this analysis includes 114 MI sessions as the unit of analysis.
Time Frame: as for outcome 2
Population: Analysis population includes the N=114 MI sessions that were completed by providers across all training groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: MI Sessions completed by providers
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
Number analyzed (MI Sessions completed by providers) | 3 | 11 | 100
score on a scale | 3.92 (0.88) | 4.25 (0.52) | 4.49 (0.46)
Statistical Analysis 1: Comparison: Do One vs Order One; Test type: Superiority; p = .1327, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.24 — Mean difference = Order One - Do One
Statistical Analysis 2: Comparison: See One vs Order One; Test type: Superiority; p = 0.4097, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.57; mean difference = Order One - See One
Statistical Analysis 3: Comparison: See One vs Do One; Test type: Superiority; p = 0.8779, Kruskal-Wallis — p-value adjusted for multiple comparisons using Dwass, Steel, Critchlow-Fligner method; Mean Difference (Final Values) = 0.33 — mean difference = Do One - See One

6. Secondary Outcome: Adequately Performing MI
Description: The Independent Tape Rater Scale includes 5 fundamental MI items and 5 advanced MI items. Items are rated for adherence on a scale of 1 (not at all) to 7 (extensively) and competency on a scale of 1 (not at all) to 7 (excellent). Higher scores are better adherence or competence. An adequately performed MI session occurs when at least half the MI consistent items are rated average or above (i.e., score of 4, 5, 6, or 7) for both adherence and competence. Percentage of MI sessions reaching this adequate performance threshold, per arm, served as the secondary outcome measure. Only MI sessions conducted within each study arm by the providers with patient participants were included in this analysis. Since 3 MI sessions were conducted by providers in See One, 11 sessions were conducted by providers in Do One, and 100 sessions were conducted by providers in Order One, this analysis includes 114 MI sessions as the unit of analysis.
Time Frame: as for outcome 2
Measure: Count of Units; unit: MI Sessions completed by providers
Units Other Than Participants: MI Sessions completed by providers
Arm/Group | See One | Do One | Order One
Number analyzed (Participants) | 13 | 12 | 13
Number analyzed (MI Sessions completed by providers) | 3 | 11 | 100
MI Sessions completed by providers | 2 | 11 | 100

ADVERSE EVENTS:
Time Frame: For provider participants, adverse events were monitored/collected over the course of their implementation trial participation from study enrollment until they were assigned their last patient participant; across provider participants, this period was up to one year. For patient participants, adverse events were monitored/collected from study enrollment through the period in which the provider participants were assigned to their care; across patient participants, this period was up to one week.
Description: The Adverse Event Table combines within each arm the number of patient participants and the number of provider participants at risk. Hence, See One includes 336 patient participants and 13 provider participants (subtotal = 349); Do One includes 379 patient participants and 12 provider participants (subtotal = 391); and Order One includes 458 patient participants and 13 provider participants (subtotal = 471). In total, we document adverse events for 1211 participants at risk.
Arm/Group | See One | Do One | Order One
All-Cause Mortality (participants affected / at risk) | 0/349 | 0/391 | 0/471
Serious Adverse Events (participants affected / at risk) | 0/349 | 0/391 | 0/471
Other Adverse Events (participants affected / at risk) | 0/349 | 0/391 | 0/471

LIMITATIONS AND CAVEATS:
This study was conducted across medical units within one urban hospital, reducing generalizability. We did not follow patients' substance use following hospital discharge; the effectiveness of MI delivered in this study is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT01825057/Prot_SAP_000.pdf